CLINICAL TRIAL: NCT03880370
Title: RELATIONSHIP OF LUMBOPELVIC MUSCULATURE WITH FUNCTIONAL TESTS IN NON-PROFESSIONAL ATHLETES WITH LUMBAR DISC HERNIATION
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Other Study IDs: 19/044-E_Tesis
Record Dates: First submitted 2019-03-04; First posted 2019-03-19 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Low Back Pain; Herniated Lumbar Disk; Sciatica
Keywords: ultrasound; functional test; herniated lumbar disk; low back pain
MeSH Terms: conditions — Low Back Pain; Sciatica | interventions — Surveys and Questionnaires; Weights and Measures; Ultrasonography; Pliability

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- group 1(group without low back pain): Participants inclusion criteria an age 18 to 55 years of age who practice sports equal to greater than three hours per week who have not had low back pain or ciatalgia in the last 12 months.
  Interventions: Behavioral: Questionnaires / scales; Diagnostic Test: Ultrasound imaging; Diagnostic Test: FLEXIBILITY; Diagnostic Test: FUNCTIONAL TESTS
- group 2 (low back pain group): Participants inclusion criteria an age 18 and 55 years of age who practice sports equal to greater than three hours a week, with a history of at least one episode of low back pain and / or ciatalgia in the last 12 months lasting no longer than three months and diagnosis of hernia lumbar disc using MRI.
  Interventions: Behavioral: Questionnaires / scales; Diagnostic Test: Ultrasound imaging; Diagnostic Test: FLEXIBILITY; Diagnostic Test: FUNCTIONAL TESTS

INTERVENTIONS:
Behavioral: Questionnaires / scales — EVA, ROLAND MORRIS, OWESTRY and Global Questionnaire of Physical Activity (GPAQ)
Diagnostic Test: Ultrasound imaging — Rectus abdominis dominant side & non-dominant side external oblique dominant side & non-dominant side internal oblique dominant side & non-dominant side transversus abdominis dominant side & non-dominant side lumbar multififidus l4-l5-s1 gluteus medius dominant side & non-dominant side
Diagnostic Test: FLEXIBILITY — weight-bearing lunge hip lateral rotation straight leg raise fingertip to floor test
Diagnostic Test: FUNCTIONAL TESTS — Star excursion balance test (sebt) prone bridging test Side bridging test Modified biering-sørensen

SUMMARY:
This is a control-case study. It has been designed to determine if there is a relationship between the cross sectional (thickness), through RUSI ultrasound, of the abdominal muscles, lumbar and hip muscles with the results of the functional tests, to determine its relevance in patients with low back pain and / or ciatalgia and lumbar disc herniation in non-professional athletes. The secondary objectives of the study will be to know if there is a relationship between the results of ultrasound measurements and functional tests with the result of the disability questionnaires, the amount of pain and its location, as well as determine the relevance, depending on the results of ultrasound measurements and test of the presence or not of a lumbar disc herniation.

ELIGIBILITY:
Inclusion criteria:

* Age 18 to 55 years of age.
* Sports practice equal to greater than three hours per week.
* No low back pain or ciatalgia in the last 12 months.

Exclusion criteria:

* Traumatic process or surgery in the lower back or lower limb in the last year.
* Alterations of the skin or local infection in the area to be examined or that impedes the ultrasonographic measurement or performance of the functional tests.
* Peripheral or central neurological pathology.
* Psychiatric pathology and / or cognitive alterations.
* Inflammatory and tumor diseases.
* Alterations that prevent the understanding of the indications and / or the performance of the tests.

Group selection criteria:

* Group 1(group without low back pain): No low back pain or ciatalgia in the last 12 months.
* Group 2 (low back pain group): History of at least one episode of low back pain and / or ciatalgia in the last 12 months lasting no longer than three months and diagnosis of hernia lumbar disc using MRI.

Ages: 18 Years to 55 Years | Sex: All
Age Groups: Adult
Study Population: Men and women between 18 and 55 years old. Non-professional sports practice equal to greater than 3 hours per week
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasound changes in muscle cross-sectional area produced of the transversus abdominis. | 5 minutes
  Ultrasound changes in muscle cross-sectional area produced of the transversus abdominis.
Ultrasound changes in muscle cross-sectional area (CSA) produced of the internal oblique. | 5 minutes
  Ultrasound changes in muscle cross-sectional area (CSA) produced of the internal oblique.
Ultrasound changes in muscle cross-sectional area (CSA)produced of the external oblique. | 5 minutes
  Ultrasound changes in muscle cross-sectional area (CSA) produced of the external oblique.
Ultrasound changes in muscle cross-sectional area (CSA)produced of the rectus abdominis. | 5 minutes
  Ultrasound changes in muscle cross-sectional area (CSA)produced of the rectus abdominis.
Ultrasound changes in muscle cross-sectional area (CSA)produced of the lumbar multifidus. | 5 minutes
  Ultrasound changes in muscle cross-sectional area (CSA)produced of the lumbar multifidus.

SECONDARY OUTCOMES:
Ultrasound changes in muscle cross-sectional area (CSA) produced of the gluteus medius. | 10 minutes
  Ultrasound changes in muscle cross-sectional area (CSA) produced of the gluteus medius.
Functional test. Star excursion balance test (SEBT) | 10 minutes
  Test Position: Standing barefoot on a grid with an anterior, posteromedial and posterolateral line at a 45° angle away from the projected anterior line.
  For the anterior test: most distal aspect of the toes aligned with the tape, centre of heel in line with the tape. For the posterior tests: most posterior aspect of the heel aligned with the tape and the second toe on the tape.
  Test: Stand barefoot with the foot aligned to the tape and hands to the side. With the other leg, reach out as far as possible in the tested direction with the most distal part of the foot. 4 practice trials are mandatory in each direction, test each direction 3 times.
  Measurement: Measure the reach distance in each direction and register the maximal reach distance in cm. The distances will be compared to each other and to the respective functional leg length. The best result is the longest distance
Functional test. Side bridging test | 10 minutes
  Test Position:
  Athlete is side-lying on an exercise mat. Both feet are in contact with the floor, the fore-arm perpendicular to the athlete's body. The other hand is holding the shoulder.
  Test:
  Athlete attains a side-bridge position, keeping both feet and one fore-arm in contact with the floor. Tester helps the athlete attain a neutral position of the lumbar spine and positions the head in the same line.
  Two practice trials are allowed. Test both sides, with at least 10 minutes of rest between sides.
  In some cases, only 1 side needs to be tested.
  Measurement:
  Measure the time the athlete is able to keep this neutral position. Correct the athlete's position if necessary, if he's unable to maintain the position for 2 consecutive seconds, stop the test. The best result is the longest time
Functional test. Modified biering-sørensen | 10 minutes
  Test Position:
  Prone position, the ASIS just over the edge of the treatment table. Arms crossed over shoulders.Neutral position of spine.
  Test:
  Instruct the athlete to maintain the neutral position as long as possible (surfaced at 4min).Test fails when the athlete is unable to maintain this position for more than 2 executive seconds (2 corrections allowed). Fail towards hyperextension/flexion. A horizontal cord at spina scapula level can be used to identify deficits.
  Measurement:
  Timing is recorded and marked in seconds. The best result is the longest time
Functional test. Prone bridging test | 10 minutes
  Test Position:
  Prone-lying with parallel forearms, thumbs up and straight legs.
  Test:
  Attain a bridging position with vertical upper arms and with the shoulder, greater trochanter and lateral malleolus in line. The head keeps in contact with an wall in front of a pacient to avoid excessive head movement. Two practice trials are allowed.
  Measurement:
  Measure the time the athlete is able to keep this frequency and the correct position. Correct the athlete's position if necessary, if he's unable to maintain the position or the frequency, stop the test. The best result is the longest time
VAS escale | 1 minute
  The most simple VAS is a straight horizontal line of fixed length, usually 100 mm. The ends are defined as the extreme limits of the parameter to be measured (symptom,pain,health) orientated from the left (worst) to the right (best).
  Scoring and Interpretation: Using a ruler, the score is determined by mea-suring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Roland-Morris Disability Questionnaire | 5 minutes
  It is used to determine the degree of disability. The extreme values oscillate between 0 (absence of disability due to low back pain) and 24 (maximum possible disability).
The Owestry Disability Index | 5 minutes
  Interpretation:
  Add the points of each section and place them in the following formula, in order to calculate your level of disability. total points / 50 X 100 =% disability (also known as: 'total points' divided by' 50 ', multiplied by' 100 = percentage of disability)
  ODI score:
  0% to 20% (minimum disability) 21% to 40% (moderate disability) 41% to 60% (severe disability) 61% to 80% (paralyzed) 81% -100%: These patients may be bedridden or may be exaggerating symptoms. A careful evaluation is recommended.
Global Questionnaire on Physical Activity (GPAQ) | 5 minutes
  The Global Physical Activity Questionnaire was developed by WHO for physical activity surveillance in countries. It collects information on physical activity participation in three settings (or domains) as well as sedentary behaviour, comprising 16 questions (P1-P16). The domains are:
  * Activity at work
  * Travel to and from places
  * Recreational activities METs (Metabolic Equivalents) are commonly used to express the intensity of physical activities, and are also used for the analysis of GPAQ data. Therefore, when calculating a person's overall energy expenditure using GPAQ data, 4 METs get assigned to the time spent in moderate activities, and 8 METs to the time spent in vigorous activities.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Plaza Manzano, Pt PhD, Principal Investigator — Universidad Complutense de Madrid

IPD SHARING:
Plan to Share IPD: No